CLINICAL TRIAL: NCT03307369
Title: A Retrospective Study to Assess the Rate of Plasmodium Vivax Infections Presenting With Severe Symptoms From 2001 to 2016 in North-western Thailand
Brief Title: A Retrospective Study of Severe Plasmodium Vivax
Acronym: SeverePV
Status: Completed | Type: Observational
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Other Study IDs: SMRU1706
Record Dates: First submitted 2017-10-05; First posted 2017-10-11 (Actual); Last update posted 2020-08-27 (Actual); Status verified 2020-08

CONDITIONS: Malaria, Vivax
Keywords: Severe malaria; plasmodium vivax
MeSH Terms: conditions — Malaria, Vivax; Malaria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Historically, Plasmodium vivax has been termed "benign" due to its non-life threatening clinical course and since the 1800's this view has been cultivated as demonstrated by the use of the term "benign tertian malaria" to describe the infection.However over the last 15 years, more severe P. vivax malaria is being reported, causing concern that severe P. vivax malaria is under diagnosed. The definition of severe P. vivax malaria borrows from P. falciparum and is primarily one of exclusion. Species PCR (polymerase chain reaction) is the only way to prove P. vivax mono-infection but is expensive and requires skilled staff and technology. In resource constrained settings, diagnostic testing is not available for detection of most non-malarial infections further affecting the ability to determine whether severe symptoms are due to P. vivax malarial infection or a concomitant one.

Retrospective studies from India, Pakistan, Indonesia, Papua New Guinea and Sudan support the existence of severe P. vivax malaria. However, inconsistent methodologies, definitions of severity, and use of diagnostic tests to exclude concomitant infection do not allow for standardised assessments for severe P. vivax infection across studies. A review by Baird, highlighted that the risk of being classed as suffering from severe illness was only minimally higher in P. falciparum than in P. vivax, but was unable to combine the data as a meta-analysis. The primary reported symptoms for severe P. vivax included severe anaemia particularly in children, severe thrombocytopaenia, respiratory distress, neurological syndromes (coma or seizures), renal and hepatic failure.

Prospective studies have shown similar results. Tjitra et al showed that 23% (675 of 2,937) patients admitted with microscopically diagnosed P. vivax infections in Papua, Indonesia had severe disease and that the risk of severe malaria was significantly higher when admitted with P. vivax than with P. falciparum. In studies from Papua New Guinea, few differences between the clinical presentation of P. falciparum and P. vivax were found in children with severe malaria. This appears to be similar in populations from Sudan, Pakistan and India. In contrast, in Thailand, anecdotal observations note a low prevalence of severe P. vivax infections.

The WHO criteria to assess severe P. falciparum have been extrapolated to P. vivax. In the 2015 WHO malaria guidelines some criteria now account for P. vivax, such as removing a minimum parasitaemia when assessing for severe anaemia. Whilst these criteria may not be the most sensitive tool to define severe P. vivax infections, it is used for this purpose. It has been suggested that additional clinical information may be necessary to define truly severe P. vivax cases.

In order to describe the characteristics of the severity of P. vivax infections in north-western Thailand, we will perform a retrospective review of annual reports of the outpatient database, the inpatient database and eligible inpatient medical records from 2001 to 2016. The WHO malaria guidelines and additional clinical information will be used to assess the severity of infection and thus, a rate of severe P. vivax can be determined.

ELIGIBILITY:
Inclusion Criteria:

* Patients voluntarily presented at SMRU clinic during 2001-2016 with a diagnosis of P. vivax mono-infection

Exclusion Criteria:

* Patients voluntarily presented at SMRU clinic during 2001-2016 with fever and were seeking consultation for the treatment of malaria or other infections.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The retrospective data from approximately 600 P.vivax infected patients who have had routine clinical work performed in the outpatient and inpatient departments at SMRU during 2001-2016. The patient population consists of refugees and migrants living along the Thailand Myanmar border in north-western Thailand who seek health care at the SMRU hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 171 (Actual)
Dates: Start 2017-10-27 (Actual); Primary Completion 2020-07-15 (Actual); Study Completion 2020-07-15 (Actual)

PRIMARY OUTCOMES:
The ratio of the number of severe cases determined to be caused by P. vivax to the number of outpatient cases treated for P. vivax | 1 year

SECONDARY OUTCOMES:
Compare the age of inpatient cases that meet or do not meet the 2015 WHO criteria for severe P. vivax | 1 year
Compare the sex of inpatient cases that meet or do not meet the 2015 WHO criteria for severe P. vivax | 1 year
Compare the medical history of inpatient cases that meet or do not meet the 2015 WHO criteria for severe P. vivax | 1 year
Compare the parasitaemia of inpatient cases that meet or do not meet the 2015 WHO criteria for severe P. vivax | 1 year
Compare the duration of hospital stay of inpatient cases that meet or do not meet the 2015 WHO criteria for severe P. vivax | 1 year
Compare the use of intravenous anti-malarial of inpatient cases that meet or do not meet the 2015 WHO criteria for severe P. vivax | 1 year
Compare the blood transfusion of inpatient cases that meet or do not meet the 2015 WHO criteria for severe P. vivax | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Shoklo Malaria Research Unit, Mae Sot, Changwat Tak, Thailand